CLINICAL TRIAL: NCT05924776
Title: Clinical Study of Plasmodium Immunotherapy for Advanced Ovarian Cancer
Brief Title: Plasmodium Immunotherapy for Advanced Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: CAS Lamvac (Guangzhou) Biomedical Technology Co., Ltd. (Industry)
Collaborators: The Third Affiliated Hospital of Southern Medical University (Other Government)
Responsible Party: Sponsor
Organization: CAS Lamvac Biotech Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFYKDX-002
Record Dates: First submitted 2023-06-19; First posted 2023-06-29 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Advanced Ovarian Cancer
Keywords: Advanced ovarian cancer; Plasmodium immunotherapy; Plasmodium vivax
MeSH Terms: conditions — Malaria, Vivax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Plasmodium immunotherapy group (Experimental): This is a single arm study that is planed to enroll 30 patients with advanced ovarian cancer and each patient will be inoculated with P.vivax-infected red blood cells containing approximately 1-5 × 10^6 Plasmodium parasites. And successful infection will be indicated by microscopic observation of parasitemia in peripheral blood samples. The treatment will last 6 weeks from the day of successful infection and will be terminated by antimalarial drugs.
  Interventions: Biological: Plasmodium immunotherapy

INTERVENTIONS:
Biological: Plasmodium immunotherapy — Inoculation 1-5 × 10^6 Plasmodium vivax once

SUMMARY:
The main purpose of this study is to evaluate the safety and effectiveness of Plasmodium immunotherapy in the treatment of advanced ovarian cancer. This study plans to enroll 30 patients with advanced ovarian cancer. Each patient is inoculated with Plasmodium vivax 1-5 × 10^6, observe the time when the parasite is detected in the peripheral blood of the subjects after the inoculation of Plasmodium, the change of the parasite density in the peripheral blood of the whole treatment cycle and the control effect of the drug on the parasite density, the main clinical symptoms and signs, laboratory test indicators, immunological test indicators and changes in the quality of life. To evaluate the safety and tolerance of the subjects to Plasmodium immunotherapy, as well as the changes of tumor related indicators and immunological indicators.

DETAILED DESCRIPTION:
Each subject who passed the screening is immunized with Plasmodium vivax 1-5 × 10^6, observe the time when the parasite is detected in the peripheral blood of the subjects after inoculation, the change of the parasite density in the peripheral blood of the whole treatment cycle (about 6 weeks) and the control effect of the drug on the parasite density. The clinical symptoms and signs after treatment are mainly observed; Blood routine, blood biochemistry, blood coagulation, tumor markers and other laboratory test indicators change; Changes of cellular immunity and humoral immunity; Changes in quality of life. When Plasmodium infected erythrocytes among total erythrocytes (defined as the parasite density) ≥ 0.1% occurs during the test, artemisinin drugs should be used to control the parasite density below 0.1%, and symptomatic treatment should be carried out. The duration of Plasmodium immunotherapy for each subject is 6 weeks (time window, ± 1 day). The day the immunodynamic marker (Fim) is greater than baseline level is defined as the first day of Plasmodium immunotherapy. When Plasmodium immunotherapy lasts for 6 weeks (time window, ± 1 day), use antimalarial drugs to kill the parasite and terminate the treatment. After treatment, the patients are followed up for 2 years. We will carry out a follow-up visit once a month after the termination of Plasmodium infection according to the plan, and the follow-up visit in the first month, third month and sixth month is outpatient visit, which is ± 5 days in the first month and ± 7 days in the third month and sixth month respectively; Follow-up outpatient visit will be conducted every 3 months ± 10 days; The rest are telephone follow-up (once every 30 days ± 5). When the follow-up time overlaps with the previous outpatient follow-up time, no additional telephone follow-up will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all the following inclusion criteria:

  1. 18-80 years old(including the threshold), female;
  2. The patients with ovarian cancer, who has been diagnosed by histopathological examination, can provide pathological reports, and is classified as stage III or stage IV according to the American Joint Committee on Cancer (AJCC) ovarian cancer staging version 8 (2017);
  3. Platinum-resistant patient who has received at least the first line of platinum-containing standard chemotherapy (refer to China's Guidelines for the Diagnosis and Treatment of Ovarian Cancer (2022)) in the past, and have been evaluated as disease progression by objective imaging;
  4. According to the evaluation standard of solid tumor efficacy RECIST 1.1, the therapeutic effect can be evaluated if there is ≥ 1 measurable lesion or continuous positive tumor marker;
  5. There are no plans and requirements for receiving other anti-tumor treatment during the treatment of Plasmodium immunotherapy;
  6. The score of Eastern Cooperative Oncology Group(ECOG) is 0-1;
  7. Expected survival time ≥ 3 months;
  8. If no platelets or red blood cells are transfused within 14 days before screening, and no thrombopoietin (TPO), granulocyte colony stimulating factor (G-CSF), granulocyte macrophage colony stimulating factor (GM-CSF), interleukin 11 (IL-11) or other drugs are used to correct abnormal blood picture: neutrophil (NEUM) ≥ 1.5 × 10^9/L, platelet (PLT) ≥ 100 × 10^9/L, hemoglobin (HGB) ≥ 90g/L, no obvious abnormality of erythrocyte morphology; Albumin (ALB) ≥ 35g/L;
  9. For female subjects with the possibility of pregnancy: from the time of signing the informed consent form (ICF) to the end of Plasmodium immunotherapy treatment at least 24 weeks, consent to abstinence or use of effective contraceptive methods, including intrauterine devices, etc. (Note: women of childbearing age have undergone surgical sterilization (including hysterectomy, bilateral oophorectomy or total hysterectomy), or have menopause for more than 24 menstrual cycles, That is, there is no possibility of pregnancy);
  10. Subjects are fully capable of understanding and signing the informed consent form.

Exclusion Criteria:

* Subjects who have any of the following conditions cannot be included in the study:

  1. Have received any investigational drug within 4 weeks before the first inoculation of Plasmodium parasite, or have participated in another clinical study at the same time (except that the subjects have participated in the observational and non-interventive clinical study, or are in the follow-up period of the intervention clinical study);
  2. Immunodeficiency diseases, including HIV infection, other acquired and congenital immunodeficiency diseases;
  3. Coagulation dysfunction, or acute or chronic hemorrhagic disease;
  4. Have received other anti-tumor treatment in the past, and the period from the termination of treatment to the screening is less than 14 days or 5 half-lives (whichever occurs first);
  5. The time interval between radiotherapy and treatment in this study for patients who have previously received external or internal radiotherapy is less than 28 days;
  6. Patients with severe hemoglobinopathy or severe Glucose-6-Phosphate Dehydrogenase(G6PD) deficiency;
  7. After splenectomy or splenomegaly;
  8. Drug addicts or alcohol addicts;
  9. Plenty of pleural effusion, pericardial effusion or ascites;
  10. Patients with active hepatitis B or hepatitis C;
  11. Patients with obvious defects in immunocyte classification test (CD4+T cell absolute count<200/ μ l）； Or receive any form of immunosuppressive treatment within 28 days before the trial treatment;
  12. Have serious or uncontrolled systemic diseases (including but not limited to active infection, grade III hypertension, unstable angina pectoris, congestive heart failure, grade III or IV heart disease, serious arrhythmia, liver and kidney insufficiency, myocardial infarction, etc.);
  13. Currently has mental disorder or a history of mental illness;
  14. Having undergone major surgery within three months from the screening period;
  15. Have received bone marrow transplantation or organ transplantation in the past;
  16. Moderate or severe pulmonary ventilation dysfunction;
  17. Those who are currently receiving regular anti-tumor treatment, and the treatment is effective or there is no obvious progress in the disease;
  18. The investigator evaluated the patients who could not tolerate Plasmodium immunotherapy;
  19. Pregnancy, lactation or pregnancy within 6 months after treatment;
  20. According to the judgment of the researcher, the other conditions of the subject are not suitable for participating in the test.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-20 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate（ORR） | 2 years
  The proportion of patients whose tumors shrink to a certain amount and remain for a certain time.
Progression-free survival (PFS) | 2 years
  Starting from treatment until the disease progression is first found or the time of any cause of death (disease progression refers to tumor growth, or metastasis of primary tumor, or discovery of new lesions).
Disease control rate (DCR) | 2 years
  The proportion of patients who had a best response rating of complete response, partial response, or stable disease.
1-year survival rate | 1 years
  The number of cancer cases remaining after 1 year of treatment / the total number of cancer cases treated * 100%.
2-year survival rate | 2 years
  The number of cancer cases remaining after 2 years of treatment / the total number of cancer cases treated * 100%.
Overall survival (OS) | 2 years
  The time starting from the treatment to death of whatever causes (when subjects have lost for follow-up before death, the last follow-up time will be calculated as the time of death).
Tumor marker level | 2 years
  The patient's sensitive tumor markers will be reviewed periodically from the time they are enrolled into the study. The tumor markers include Carcinoembryonic antigen（CEA）, Carbohydrate Antigen 125（CA125）, human epididymis protein 4（HE4）, alpha-fetal protein（AFP）, neuron-specific enolase（NSE）, Carbohydrate Antigen 199（CA199）.

SECONDARY OUTCOMES:
Incidence of adverse events (AE) and serious adverse events (SAE) | 2 years
  Any adverse medical event occurred in the subjects who participated in the clinical study and received Plasmodium immunotherapy.
Pain score | 2 years
  Patients are regularly evaluated with Visual Analog Scale for Pain. The minimum value is 0, and the maximum value is 10. The higher scores mean a worse outcome.

OTHER OUTCOMES:
Immunological indicators | 2 years
  Detection of absolute number of immune cells（such as CD3+CD4+、CD3+CD8+ and so on）in peripheral blood by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Guo Shuiqun, Ph.D., M.D., Principal Investigator — The Third Affiliated Hospital of Southern Medical University
Locations (1):
- The Third Affiliated Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No